CLINICAL TRIAL: NCT03954704
Title: A Phase 1a/1b Study of GS-1423, an Anti-CD73-TGFβ-Trap Bifunctional Antibody, as Monotherapy or in Combination With a Chemotherapy Regimen in Subjects With Advanced Solid Tumors
Brief Title: Study of Dalutrafusp Alfa (Formerly GS-1423) in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to discontinue the study was made based on the totality of the clinical, pharmacokinetic, and pharmacodynamic findings. No safety concerns were observed.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-505-5452; 2019-004938-41 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a, Part A - Dose Escalation (Experimental): Part A will consist of dose escalation by an accelerated dosing design and a 3+3 dose escalation scheme. Participants will receive escalating dose levels dalutrafusp alfa of up to 45 mg/kg on Day 1 of each 2-week cycle (Q2W) until the participant meets study treatment discontinuation criteria or for up to 1 year.
  Interventions: Drug: Dalutrafusp alfa
- Phase 1a, Part B - Flat Dose Regimen (Experimental): Part B will consist of 3 adaptive cohorts. Based on PK, pharmacodynamics, and safety results from the Part A study, participants will be administered a flat dose of dalutrafusp alfa on Day 1 of each cycle QW, Q2W and/or every 3 weeks (Q3W) until the participant meets study treatment discontinuation criteria or for up to 1 year.
  Interventions: Drug: Dalutrafusp alfa
- Phase 1b, Cohort 1 (Gastric Cancer) (Experimental): Safety run-in: A standard 3+3 dose escalation design will be used to determine the DLT and MTD or RP2D of dalutrafusp alfa in combination with mFOLFOX6. The planned starting dose of dalutrafusp alfa will be targeted to achieve the exposure at -1 dose of RP2D monotherapy (Q2W) determined from Phase 1a. Dalutrafusp alfa will be administered in combination with mFOLFOX6.
  Post safety run-in: Approximately 70 participants will be enrolled to receive dalutrafusp alfa at the dose level determined from the safety run-in period, in combination with mFOLFOX6 regimen.
  Participants will receive dalutrafusp alfa on Day 1 of each 14-day cycle up to 2 years until PD, or unacceptable toxicity, substantial noncompliance with study procedures or study drug, study discontinuation or withdrawal from study. Participants will also receive mFOLFOX6 regimen Q2W for up to 12 cycles.
  Interventions: Drug: Dalutrafusp alfa; Drug: mFOLFOX6 Regimen
- Phase 1b, Cohort 2 (Paired Biopsy) (Experimental): Participants will receive dalutrafusp alfa at the dose level determined from Phase 1a Q2W until the participants meets study treatment discontinuation criteria or for up to 1 year.
  Interventions: Drug: Dalutrafusp alfa

INTERVENTIONS:
Drug: Dalutrafusp alfa — Administered intravenously
  Other Names: GS-1423
  Arms: Phase 1a, Part A - Dose Escalation; Phase 1b, Cohort 1 (Gastric Cancer); Phase 1b, Cohort 2 (Paired Biopsy)
Drug: mFOLFOX6 Regimen — Chemotherapy regimen of oxaliplatin, 5-fluorouracil [5-FU], and leucovorin
  Arms: Phase 1b, Cohort 1 (Gastric Cancer)
Drug: Dalutrafusp alfa — Administered intravenously
  Other Names: GS-1423
  Arms: Phase 1a, Part B - Flat Dose Regimen

SUMMARY:
For Phase 1a Part A, the primary objectives are to assess safety and tolerability and to define the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of dalutrafusp alfa (formerly GS-1423) monotherapy in participants with advanced solid tumors.

For Phase 1a Part B, the primary objective is to assess safety and tolerability of dalutrafusp alfa monotherapy in participants with advanced solid tumors.

For Phase 1b Cohort 1 safety run-in, the primary objective is to assess safety and tolerability and to define the DLT and MTD or RP2D of dalutrafusp alfa in combination with a chemotherapy regimen in participants with advanced gastric or gastroesophageal junction adenocarcinoma.

For Phase 1b Cohort 1 post safety run-in, the primary objective is to assess the preliminary efficacy of dalutrafusp alfa in combination with a chemotherapy regimen in participants with advanced gastric or gastroesophageal junction adenocarcinoma, as assessed by the confirmed objective response rate (ORR).

For Phase 1b Cohort 2, the primary objective is to assess safety and tolerability of dalutrafusp alfa monotherapy in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis:

  * For Phase 1a and Phase 1b Cohort 2, have a histologically or cytologically confirmed diagnosis of a locally advanced or metastatic solid tumor for which no standard therapy is available (per local guidance) or standard therapy has failed, or
  * For Phase 1b Cohort 1, have histologically or cytologically confirmed unresectable, recurrent or metastatic gastric or gastroesophageal junction adenocarcinoma who have not previously received systemic therapy for advanced disease
* Measurable disease: Have measurable disease on imaging based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
* Have a life expectancy of at least 3 months and an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Key Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 3 weeks of the first dose of treatment
* Has persisting toxicity related to prior therapy of National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE) Grade >1 severity
* Is expected to require any other form of systemic or localized anticancer therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection)
* Has concurrent active malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix or superficial bladder cancer who has undergone potentially curative therapy with no evidence of disease. Individuals with other previous malignancies are eligible if disease-free for >2 years
* Has a known central nervous system metastasis(es), unless metastases are treated and stable and the individual does not require systemic corticosteroids for management of CNS symptoms at least 7 days prior to study treatment. Individuals with history of carcinomatous meningitis are excluded regardless of clinical stability.
* Has active or history of autoimmune disease that has required systemic treatment within 2 years of the start of trial treatment

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - Scottsdale Healthcare Hospitals d/b/a HonorHealth, Scottsdale, Arizona
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tolcher AW, Gordon M, Mahoney KM, Seto A, Zavodovskaya M, Hsueh CH, Zhai S, Tarnowski T, Jurgensmeier JM, Stinson S, Othman AA, Chen T, Strauss J. Phase 1 first-in-human study of dalutrafusp alfa, an anti-CD73-TGF-beta-trap bifunctional antibody, in patients with advanced solid tumors. J Immunother Cancer. 2023 Feb;11(2):e005267. doi: 10.1136/jitc-2022-005267. PMID 36746510
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-505-5452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 03 June 2019. The last study visit occurred on 15 April 2021.
Pre-assignment Details: The study was discontinued prior to initiation of Phase 1a Part B and Phase 1b. Therefore, data are reported for only Phase 1a Part A.
Groups:
- Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg: GS-1423 0.3 mg/kg of body weight, solution for intravenous (IV) infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg: GS-1423 1 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg: GS-1423 3 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg: GS-1423 10 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg: GS-1423 20 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg: GS-1423 30 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg: GS-1423 45 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
Period: Overall Study
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Started | 1 | 1 | 3 | 3 | 3 | 8 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 3 | 8 | 3
Not completed — Death | 1 | 1 | 1 | 3 | 2 | 2 | 0
Not completed — Withdrew Consent | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0 | 1 | 4 | 2
Not completed — Enrolled but not Treated | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg: GS-1423 0.3 mg/kg of body weight, solution for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
- Total: Total of all reporting groups
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 | 67 | 70 (8.7) | 70 (11.6) | 62 (7.4) | 57 (15.8) | 71 (7.2) | 64 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 2 | 2 | 6 | 1 | 15
  Male | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 3 | 2 | 5 | 2 | 14
  Not Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
  White | 1 | 1 | 3 | 3 | 2 | 5 | 3 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a Part A: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs), Graded Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0)
Description: DLT was defined as: Grade 3 thrombocytopenia with bleeding; Grade ≥ 3 febrile neutropenia; any Grade 4 hematologic laboratory abnormalities/adverse events (AEs) (except Grade 4 lymphopenia and anaemia, Grade 4 neutropenia lasting ≤ 7 days with no fever); Grade 4 non-hematologic AEs; any ≥Grade 2 uveitis, blurred vision, eye pain, and/or reduction of visual acuity that did not respond to topical therapy and did not improve to Grade 1 severity within 2 weeks of topical therapy initiation or required systemic treatment; Grade 3 non-hematologic AEs; any other non-immune-related Grade 3 AE (except any Grade 3 endocrinopathy; Grade 3 AE of tumor flare; transient [≤ 3 days] Grade 3 fatigue, local reactions, headache, nausea, emesis, or diarrhea and/or resolved to Grade ≤ 1; transient Grade 3 flu-like symptoms or fever); inability to receive first 2 doses of GS-1423 or > 2-week delay in starting next cycle of therapy due to a treatment-related toxicity; Grade 5 event (death).
Time Frame: Baseline up to 28 days
Population: The DLT-Evaluable Analysis Set included all participants who were enrolled for dose escalation, received the protocol-specified treatment, and completed safety procedures through Day 28 (inclusive) or experienced a DLT prior to Day 28.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 5 | 3
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Phase 1a Part A: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant administered the study drug, which did not necessarily have a causal relationship with the treatment. An AE could therefore, be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Adverse events might also include pretreatment or posttreatment complications that occurred as a result of protocol-specified procedures or special situations. Preexisting events that increased in severity or change in nature during or as a consequence of participation in the study were also considered AEs. TEAEs were AEs with onset dates on or after the first dose of study drug GS-1423 and up to 30 days after permanent withdrawal of GS-1423.
Time Frame: First dose date up to permanent withdrawal of GS-1423 (maximum duration: 26.3 weeks) plus 30 days
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 3
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

3. Secondary Outcome: Phase 1a Part A: Percentage of Participants With Treatment-Emergent Grade 3 or 4 Laboratory Abnormalities
Description: Severity was graded per NCI CTCAE v5.0. Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening or disabling, Grade 5: Death related to AE.
Time Frame: First dose date up to permanent withdrawal of GS-1423 (maximum duration: 26.3 weeks) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg: GS-1423 3 mg/kg solution of body weight, for IV infusion, administered over approximately 60 minutes, on Day 1 of each 2-week cycle until the participant met study treatment discontinuation criteria or for up to 1 year.
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 3
percentage of participants
  Hematology | 0 | 100.0 | 0 | 0 | 33.3 | 14.3 | 0
  Serum Chemistry | 0 | 0 | 0 | 33.3 | 33.3 | 14.3 | 0
  Coagulation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Endocrine Function Tests | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Phase 1a Part A: Percentage of Participants With Shift in Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG) From Baseline to Overall Study
Description: The Baseline value was the last available value collected on or prior to first dose of study drug. Percentages were based on participants with values available at both baseline and postbaseline.
  NCS = Non-clinical significance; CS = Clinical significance.
Time Frame: First dose date up to permanent withdrawal of GS-1423 (maximum duration: 26.3 weeks) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 3
percentage of participants
  Normal baseline - Normal | 0 | 0 | 33.3 | 33.3 | 0 | 0 | 0
  Normal baseline - Abnormal NCS | 0 | 0 | 0 | 33.3 | 66.7 | 71.4 | 0
  Normal baseline - Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS Baseline - Normal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS Baseline - Abnormal NCS | 100.0 | 100.0 | 66.7 | 33.3 | 33.3 | 28.6 | 100.0
  Abnormal NCS Baseline - Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal CS Baseline - Normal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal CS Baseline - Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal CS Baseline - Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Phase 1a Part A: Pharmacokinetic (PK) Parameter: AUCtau of GS-1423
Description: AUCtau was defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Cycle 1 and Cycle 4: Day 1 (Predose, end of infusion, 2 and 6 hours post start of infusion); Days 2, 3, 5, and 8 (additionally at Day 15 in Cycle 4)
Population: Participants in the PK Analysis Set (all enrolled participants who received at least 1 dose of study drug and had at least 1 non-missing postdose concentration value reported by the PK laboratory) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Number analyzed (Participants) | 0 | 0 | 3 | 3 | 3 | 6 | 3
µg*h/mL
  Cycle 1 |  |  | 1476.9 (759.84) | 5311.8 (595.77) | 33530.9 (1646.22) | 51593.2 (16313.20) | 64856.3 (9814.95)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 3 | 0 | 1 | 2 | 1
  Cycle 4 |  |  | 1711.9 (1486.08) |  | 28558.0 | 65368.1 (5469.82) | 74097.0

6. Secondary Outcome: Phase 1a Part A: Percentage of Participants Who Developed Anti-Drug Antibodies (ADAs)
Time Frame: Baseline, during the treatment (maximum duration: 26.3 weeks), Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 4 Day 15, Cycle 6 Day 1, 30-day follow-up (30 days after discontinuation of GS-1423), post treatment follow-up (3 months)
Population: The Immunogenicity Analysis Set included all participants in the Safety Analysis Set who have at least 1 nonmissing postdose ADA status reported.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 3
percentage of participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 14.3 | 0
  During the Treatment | 100.0 | 0 | 66.7 | 66.7 | 66.7 | 0 | 33.3
  Cycle 2 Day 1 | 0 | 0 | 0 | 66.7 | 33.3 | 0 | 33.3
  Cycle 3 Day 1 | 0 | 0 | 33.3 | 33.3 | 66.7 | 0 | 0
  Cycle 4 Day 1 | 0 | 0 | 33.3 | 0 | 33.3 | 0 | 0
  Cycle 4 Day 15 | 0 | 0 | 0 | 0 | 33.3 | 0 | 0
  Cycle 6 Day 1 | 0 | 0 | 33.3 | 0 | 0 | 0 | 0
  30-Day Follow-Up | 100.0 | 0 | 0 | 0 | 33.3 | 0 | 0
  Post Treatment Follow-Up (3 months) | 0 | 0 | 0 | 0 | 33.0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: First dose date up to 30 days after permanent withdrawal of GS-1423 (maximum exposure: 26.3 weeks); All-Cause Mortality: Enrollment up to 22 months
Description: Adverse Events and Serious Adverse Events: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
  All-Cause Mortality: All Enrolled Analysis Set included all participants who received a study participant identification number in the study after screening.
Arm/Group | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/3 | 3/3 | 2/3 | 2/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/3 | 2/3 | 2/3 | 4/7 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 3/3 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg (N=1) | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg (N=1) | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg (N=3) | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg (N=3) | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg (N=3) | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg (N=7) | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic embolus (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a (Part A) Cohort 1: GS-1423 0.3 mg/kg (N=1) | Phase 1a (Part A) Cohort 2: GS-1423 1 mg/kg (N=1) | Phase 1a (Part A) Cohort 3: GS-1423 3 mg/kg (N=3) | Phase 1a (Part A) Cohort 4: GS-1423 10 mg/kg (N=3) | Phase 1a (Part A) Cohort 5: GS-1423 20 mg/kg (N=3) | Phase 1a (Part A) Cohort 6: GS-1423 30 mg/kg (N=7) | Phase 1a (Part A) Cohort 7: GS-1423 45 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 2 | 4 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Because the study was terminated after enrolling only 22 participants in the dose-escalation stage (Phase 1a Part A), planned analysis was not conducted for Phase 1a Part B, and Phase 1b.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT03954704/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03954704/SAP_001.pdf